CLINICAL TRIAL: NCT00806078
Title: A Comparison of the Bioavailability of Quinine Sulfate Capsules Following a 648 mg Dose When Mixed in Chocolate Pudding Relative to That With Intact Capsules in Healthy Adults Under Fasting Conditions
Brief Title: Comparison Bioavailability Study of Quinine Sulfate in Chocolate Pudding
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-07-1004
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Healthy; Bioequivalence; Pharmacokinetics
MeSH Terms: interventions — Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single dose intact capsules 2 x 324 mg
  Interventions: Drug: quinine sulfate
- 2 (Experimental): Single dose contents of two capsules (2 x 324 mg) opened and mixed in 120 mL of chocolate pudding
  Interventions: Drug: quinine sulfate

INTERVENTIONS:
Drug: quinine sulfate — 2 x 324 mg capsules (648 mg)
  Other Names: Qualaquin
  Arms: 1
Drug: quinine sulfate — 2 x 324 mg capsules (648 mg)
  Other Names: Qualaquin
  Arms: 2

SUMMARY:
This is an open label randomized single dose two-way crossover study to compare the bioavailability of a single oral dose of quinine sulfate 648 mg(2 x 324 mg) when mixed with 120 ml of chocolate pudding relative to the same dose given as two intact capsules.

DETAILED DESCRIPTION:
Prior studies have shown that intact quinine sulfate capsules can be taken without regard for food. This is an open label randomized single dose two-way crossover study to compare the bioavailability of a single oral dose of quinine sulfate 648mg(2 x 324 mg capsules) when opened and mixed with 120 ml of chocolate pudding relative to the same dose given as two intact capsules. Eighteen healthy adult subjects will be enrolled. Following a fast of at least 10 hours subjects will be randomized to receive either 648 mg of quinine sulfate as the intact capsules or opened mixed in 120ml of chocolate pudding. Following a washout period of at least 7 days all subjects will be given the alternate dose under similar conditions. Following each dose, blood samples will be collected at times sufficient to determine the difference in bioavailability (if any) between the two methods of drug administration. In addition patients will be monitored for any adverse events including Electrocardiogram (EKG) changes (at baseline and 4 hours after each dose).

ELIGIBILITY:
Inclusion Criteria:

* Healthy nonsmoking adults with hemoglobin at least 12 g/dl. Males at least 52 kg, females at least 45kg with body mass index in the normal range, females must be chemically or surgically sterile or postmenopausal (amenorrhea at least 2years)

Exclusion Criteria:

* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) Recent (1-year) history or evidence of alcoholism or drug abuse History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease, myasthenia gravis, optic neuritis or Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Prolonged corrected QT interval(QTc) on Electrocardiogram(EKG) at screening -males >430 msec, females >450 msec.

PR interval on EKG >200 msec at screening or prior to dose in either dosing period

* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 30 days prior to the first dose and throughout the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, MD, Principal Investigator — MDS Pharma Services; Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- MDS Pharma Services, Saint Laurent, Montreal, Quebec, Canada

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.HTML
- See also: Daily Med — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive a single dose of quinine 648 mg (2 x 324 mg) either as intact capsules or capsules opened and their contents mixed in 120 mL chocolate pudding after a fast of at least 10 hours. Following a 7 day wash out period, all participants were given the alternate dose under similar conditions.
Groups:
- Quinine Alone First: Participants were randomized to receive a single dose of quinine 648 mg (2 x 324 mg) as intact capsules after a fast of at least 10 hours. Blood was drawn at times sufficient to characterize quinine pharmacokinetics after this dose. Following a 7 day wash out period, all participants were given quinine 648 mg (2 x 324 mg) as capsules opened and their contents mixed in 120 mL chocolate pudding under similar conditions.
- Quinine With Chocolate Pudding First: Participants were randomized to receive a single dose of Quinine 648 mg (2 x 324 mg capsules) opened and mixed in 120 mL chocolate pudding after a fast of at least 10 hours. Blood was drawn at times sufficient to characterize the pharmacokinetics of quinine after this dose. Following a 7 day wash out period, all participants were given Quinine 648 mg (2 x 324 mg) as intact capsules under similar conditions.
Period: First Intervention
Arm/Group | Quinine Alone First | Quinine With Chocolate Pudding First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: 7 Day Washout Period
Arm/Group | Quinine Alone First | Quinine With Chocolate Pudding First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Quinine Alone First | Quinine With Chocolate Pudding First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Quinine Alone First: After a fast of at least 10 hours, participants received a single dose of quinine 648 mg (2 x 324 mg) as intact capsules. Blood was drawn sufficient to characterize the pharmacokinetics of quinine after this dose.
- Quinine With Chocolate Pudding First: After a fast of at least 10 hours participants received a single dose of quinine 648 mg (2 x 324 mg) capsules opened and mixed in 120 mL chocolate pudding. Blood was drawn at times sufficient to characterize the pharmacokinetics of quinine after this dose.
- Total: Total of all reporting groups
Arm/Group | Quinine Alone First | Quinine With Chocolate Pudding First | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.4) | 35.5 (8.4) | 35.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The highest concentration of drug in plasma after a dose. Measured to evaluate the bioequivalence of the two dosing methods
Time Frame: After dosing at time points 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, and 48 hours
Population: Analysis was performed per protocol
Measure: Mean (Standard Deviation); unit: ng per mL
Groups:
- Quinine Alone: After a fast of at least 10 hours, participants received a single dose of quinine 648 mg (2 x 324 mg) as intact capsules. Blood was drawn sufficient to characterize the pharmacokinetics of quinine after this dose.
- Quinine With Chocolate Pudding: After a fast of at least 10 hours participants received a single dose of quinine 648 mg (2 x 324 mg) capsules opened and mixed in 120 mL chocolate pudding. Blood was drawn at times sufficient to characterize the pharmacokinetics of quinine after this dose.
Arm/Group | Quinine Alone | Quinine With Chocolate Pudding
Number analyzed (Participants) | 18 | 18
ng per mL | 3291.411 (658.529) | 3439.867 (646.818)

2. Primary Outcome: Area Under the Concentration Time Curve From Zero to t. (AUC 0-t)
Description: The area under the plasma concentration versus time curve from zero to the last measurable plasma concentration as calculated by the linear trapezoidal method. Calculated to determine whether the 2 methods of administration are bioequivalent.
Time Frame: After dosing at time points 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, and 48 hours
Population: Analysis was performed per protocol
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Quinine Alone | Quinine With Chocolate Pudding
Number analyzed (Participants) | 18 | 18
ng·h/mL | 555973.3 (15455.81) | 56008.6 (12979.18)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity. (AUC Inf)
Description: AUC inf is calculated as the sum of the AUC 0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.It is calculated to evaluate the bioequivalence of the two dosing methods
Time Frame: After dosing at time points 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, and 48 hours
Population: Analysis was performed per protocol
Measure: Mean (Standard Deviation); unit: ng-h/ml
Arm/Group | Quinine Alone | Quinine With Chocolate Pudding
Number analyzed (Participants) | 18 | 18
ng-h/ml | 61887.4 (18880.15) | 60764.9 (14998.61)

ADVERSE EVENTS:
Arm/Group | Quinine Alone First | Quinine With Chocolate Pudding First
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinine Alone First (N=18) | Quinine With Chocolate Pudding First (N=18)
Feeling hot (General disorders) | 3 (5) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days